CLINICAL TRIAL: NCT01600664
Title: Randomized Controlled Trial to Evaluate the Effect of 3 Months Use With Interactive Computer Game- "My Diabetic Friend"-Comparing to Conventional Diabetes Education on Metabolic Control, Quality of Life and Diabetes Knowledge in Children With Type 1 Diabetes.
Brief Title: The Effect of the Use of Computer Game- "My Diabetic Friend" in Children With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Intel Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: rmc006814ctil
Record Dates: First submitted 2012-05-16; First posted 2012-05-17 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; "My Diabetic friend"; interactive computer game
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- interactive computer game (Experimental): Participants will be using the interactive computer game- "My Diabetic Friend", installed on Intel-powered convertible classmate PC.
  Interventions: Behavioral: Interactive computer game
- Convertible PC (Active Comparator): Participants will be using the convertible classmate PC without the interactive computer game
  Interventions: Behavioral: Convertible PC

INTERVENTIONS:
Behavioral: Interactive computer game — Participants will use the interactive computer game installed on a convertible PC
  Arms: interactive computer game
Behavioral: Convertible PC — Participants will be using the convertible PC without the interactive computer game
  Arms: Convertible PC

SUMMARY:
A randomized controlled study to evaluate the effect of 3 months use with interactive computer game- "My Diabetic Friend"- comparing to conventional diabetes education on metabolic control, quality of life and diabetes knowledge.Patients will be randomized into two groups- one group will be supplied with interactive computer game, "My Diabetic friend", installed on a computer designed for children's educational needs for a period of three months and the other group will be supplied with the same computer without the interactive computer game for three months. Metabolic control, quality of life and diabetes knowledge will be evaluated before and after the use of the computer.

The trial is consisting of two main periods: 3 months of the main study period and an optional extension period consisting of the following 3 months :

The study will include two main periods;

1. Period 1 which will last 3 months, in a randomized controlled manner, this period will serve as the main study period to assess the primary and secondary endpoints of the study.
2. Period 2: this extension period will not be an integral part of the study, and only patients who are willing will take part at this period, will continue to participate at the optional extension period. During the extension period, patients in the intervention group will be offered to continue the use of the Computer game -"My diabetic friend) for the following 3 months, and patients who participated at the control group during period 1, will be offered to start to use the Computer Game - "My Diabetic Friend" for the following 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes diagnosed at least one year prior to study entry.
2. Age:7-11 years old.
3. Treatment either with CSII or MDI.
4. HbA1c>8.0%
5. Signing an informed consent form.

Exclusion Criteria:

1. Any significant disease or conditions, including psychiatric disorders that in the opinion of the investigator are likely to affect subject compliance or subject's ability to complete the study.
2. Inability to understand/ complete the questionnaires.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Quality of life | After 12 weeks (end of study)
  Quality of life questionnaires will be completed

SECONDARY OUTCOMES:
Metabolic control | After 12 weeks (end of study)
  HbA1c will be measured
Diabetes knowledge | After 12 weeks
  Diabetes knowledge questionnaires will be completed
Patient's gaming duration | After 12 weeks
  The frequency and the duration of use of the interactive computer game by each participant will be monitored by the study team
Compliance to diabetes treatment | After 12 weeks
  Patient's parents will undergo clinical interview about patient's diabetes adherence
Average glucose levels | After 12 weeks (end of study)
Average number of blood glucose measurements | After 12 weeks (end of study)
Measurements within normal range | After 12 weeks (end of study)
Hypoglycemia events | After 12 weeks (end of study)
Hyperglycemia events | After 12 weeks (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, Principal Investigator — Rabin Medical Center
Locations (1):
- Schneider Medical Center, Petah Tikva, Israel